CLINICAL TRIAL: NCT00514878
Title: Development of a Predictive Model for Post-Discharge Nausea and Vomiting (PDNV)
Acronym: Apfel-PDNV
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Christian C. Apfel, MD, PhD, University of California
Other Study IDs: H54427-30684
Record Dates: First submitted 2007-08-08; First posted 2007-08-10 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2008-12

CONDITIONS: Nausea; Postoperative Nausea and Vomiting; Postdischarge Nausea and Vomiting; Postoperative Pain
Keywords: nausea; postoperative nausea and vomiting; postoperative pain
MeSH Terms: conditions — Nausea; Postoperative Nausea and Vomiting; Vomiting; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Adult same-day outpatients scheduled for general anesthesia

SUMMARY:
The primary purpose of this prospective cohort study is to develop a simplified risk model for post-discharge nausea and vomiting (PDNV) in adult same-day surgery patients in the US that will allow clinicians to identify those patients who would benefit from prophylactic antiemetic strategies.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* scheduled for an elective outpatient surgical procedure
* understands the nature and purpose of this survey and has signed an informed consent form
* willing and able to complete daily components of the Patient Diary from the day of surgery until the end of the 48 hour assessment
* undergoing general anesthesia requiring a tracheal tube or laryngeal mask airway

Exclusion Criteria:

* planned inpatient surgery
* inability to communicate in English
* regional anesthesia alone without general anesthesia, as PONV in this setting is known to be significantly lower [18, 19]
* persistent or recurrent nausea and/or vomiting before anesthesia due to other etiologies, unless clearly related only to the anxiety due to impending surgery
* minors (< 18 years of age)
* current pregnancy by self-report (potentially confounding for etiology of nausea)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for elective outpatient surgery
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian C Apfel, MD, PhD, Study Director — Perioperative Clinical Research Core, University of California San Francisco
Locations (1):
- Perioperative Clinical Research Core, University of California, San Francisco, California, United States